CLINICAL TRIAL: NCT05002140
Title: A Phase 1, Open-Label, Dose-Finding, Pharmacokinetic, and Pharmacodynamic Study of XRD-0394 in Subjects With Metastatic, Locally Advanced, or Recurrent Cancer Receiving Palliative Radiotherapy
Brief Title: Trial of XRD-0394, a Kinase Inhibitor, in Combination With Palliative Radiotherapy in Advanced Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: XRad Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: X0394-001
Record Dates: First submitted 2021-07-11; First posted 2021-08-12 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Metastasis; Locally Advanced Solid Tumor; Recurrent Cancer
Keywords: Ataxia telangiectasia mutated kinase; ATM; DNA-PK; DNA-dependent protein kinase; Dual inhibitor; Cancer; Palliative radiotherapy; Single dose
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- XRD-0394 40 mg (Experimental): Subjects will receive a single dose of XRD-0394 capsules approximately 90 minutes before RT on Day 2 of the RT regimen
  Interventions: Drug: XRD-0394; Radiation: Palliative radiotherapy
- XRD-0394 80 mg (Experimental): Subjects will receive a single dose of XRD-0394 capsules approximately 90 minutes before RT on Day 2 of the RT regimen
  Interventions: Drug: XRD-0394; Radiation: Palliative radiotherapy
- XRD-0394 160 mg (Experimental): Subjects will receive a single dose of XRD-0394 capsules approximately 90 minutes before RT on Day 2 of the RT regimen
  Interventions: Drug: XRD-0394; Radiation: Palliative radiotherapy
- XRD-0394 (Dose TBD) (Experimental): Subjects will receive a single dose of XRD-0394 capsules approximately 90 minutes before RT. A single biopsy will be performed in each subject (either after RT alone or after XRD-0394 and RT).
  Interventions: Drug: XRD-0394; Radiation: Palliative radiotherapy

INTERVENTIONS:
Drug: XRD-0394 — Single ascending dose
Radiation: Palliative radiotherapy — 4 Gy × 5 daily fractions

SUMMARY:
XRD-0394 is a novel, potent, oral, small molecule dual inhibitor of ataxia telangiectasia mutated kinase (ATM) and deoxyribonucleic acid (DNA)-dependent protein kinase (DNA-PK) that has selectivity compared with other phosphatidylinositol 3-kinase-related kinase (PIKK) family enzymes. This is a first-time-in-human study, which means that it is the first time the study drug is being used in humans. The purpose of the study is to evaluate the safety and tolerability of single doses of XRD-0394 administered with palliative radiotherapy (RT) to subjects with metastatic, locally advanced, or recurrent cancer. The pharmacokinetic (PK) profile and pharmacodynamic (PD) effects of single-dose XRD-0394 administered in combination with palliative RT will also be characterized.

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, open-label, dose-finding, PK and PD study of XRD-0394 in subjects with metastatic, locally advanced, or recurrent cancer receiving palliative RT. The study will evaluate single-dose PK of XRD-0394 administered to serial cohorts of subjects with the intent of identifying an oral dose that achieves plasma drug concentrations within a specified therapeutic range. Once target plasma concentrations of XRD-0394 are reached, one or more PD cohorts of subjects will be enrolled in order to demonstrate inhibition of radiation-induced ATM activity in tumor biopsy samples from subjects who received the selected dose(s).

Single Dose Escalation: Eligible subjects will be enrolled in serial cohorts to evaluate the PK of single ascending doses of XRD-0394. Dose escalation of XRD-0394 will proceed based on a standard 3+3 design. The starting dose of XRD-0394 will be 40 mg, followed by planned doses of 80 mg and 160 mg. Following administration of a single-dose of XRD-0394 and completion of RT, subjects will be evaluated for the occurrence of dose-limiting toxicities (DLTs). The available PK and safety data for each cohort will be reviewed at the conclusion of the DLT evaluation period before the decision to escalate to the next dose is made. The evaluation of additional doses of XRD-0394 will be determined based on the safety and PK data collected at completed dose levels. Dose escalation may continue until the objectives of the study are met and/or the maximum tolerated dose (MTD) of XRD-0394 is reached. PK samples for measurement of plasma concentrations of XRD-0394 will be collected pre-dose and at specified time points following XRD-0394 administration. Safety and tolerability of each XRD-0394 dose level will be evaluated by assessment of treatment-emergent adverse events (TEAEs), DLTs, and discontinuations due to TEAEs. A Safety Monitoring Committee (SMC) will be used during the study to monitor subject safety and evaluate potential DLTs.

Pharmacodynamic Assessment: The dose identified to produce plasma drug concentrations of XRD-0394 within a targeted therapeutic range will be further evaluated in separate PD cohort(s) of subjects. Subjects enrolled in a PD cohort must have a target tumor with a soft tissue component that is accessible for biopsy and must agree to undergo 1 biopsy during their RT regimen. PK samples for measurement of plasma concentrations of XRD-0394 will be collected from all subjects at pre-dose and at specified time points after XRD-0394 administration. Safety and tolerability of XRD-0394 will be evaluated by assessment of TEAEs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of cancer with clear evidence of metastasis on imaging. Subjects with locally advanced or recurrent (non-metastatic) cancer for whom palliative RT is indicated may also be enrolled.
* Scheduled to receive palliative RT delivered as 4 Gray × 5 daily fractions at the discretion of the treating radiation oncologist. The radiation plan should be designed to optimally limit the radiation dose delivered to normal tissues using conformal treatment plans and protocol-specified limits.
* One or more of the following sites of metastasis:

  * Skin
  * Subcutaneous or soft tissue
  * Any other site that will allow the radiation dose to normal structures to remain within protocol-specified dosing limits.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Male or female subjects at least 18 years of age who are willing and able to provide written informed consent.
* Other protocol-defined criteria may apply

Exclusion Criteria:

* Prior radiotherapy to the same region within the last 6 months.
* Subjects who are currently receiving palliative RT for brain metastases. Subjects who have brain metastases may participate in this trial, if they are receiving palliative RT for cancer in a location other than the brain.
* For subjects with cancers involving the spinal cord, the length of the spinal cord requiring palliative treatment must be 10 cm or less.
* Subjects with bone marrow impairment as evidenced by hemoglobin <8.0 g/dL, neutrophil count <0.7 × 10^9/L, or platelets <80 × 10^9/L .
* History of difficulty swallowing, malabsorption or other chronic gastrointestinal disease or condition that may hamper compliance and/or absorption of XRD-0394, use of percutaneous endoscopic gastrostomy (PEG) tubes.
* Significant cardiac conduction abnormalities, including a history of long corrected QT (QTc) interval syndrome and/or pacemaker, or impaired cardiovascular function such as New York Heart Association classification >2.
* Chemotherapy, immunotherapy, hormonal therapy, biologic therapy, or any other anticancer therapy within 14 days of first XRD-0394 dose. These treatments should also be held for a minimum of 14 days after completion of RT.
* Subjects receiving bleomycin within 30 days of the first dose of XRD-0394.
* Subjects receiving treatment with any drug that is a strong inhibitor or inducer of cytochrome P450 (CYP) 3A4 enzyme activity or an inhibitor of breast cancer resistance protein (BCRP) within 14 days or 5 half-lives prior to screening (whichever is longer). In particular,

  * Glucocorticoids are inducers of CYP3A4. Therefore, dexamethasone, prednisone, or other glucocorticoids should not be administered within 14 days or 5 half-lives prior to screening (whichever is longer) and should only be initiated after the course of palliative RT is complete (and at least 24 hours after the administration of XRD-0394).
  * Gefitinib and imatinib are inhibitors of BCRP. Therefore, these agents should not be administered within 14 days or 5 half-lives prior to screening (whichever is longer) and should be held for a minimum of 14 days after completion of RT.
* Participation in another investigational study of an unapproved drug or device or treatment with another ATM, DNA-PK, or ataxia-telangiectasia and Rad3-related (ATR) inhibitor within 28 days of the first dose of XRD-0394.
* Subjects who are pregnant or breast-feeding.
* Subjects with a QTc interval >450 msec (calculated using Fridericia's QT correction formula) at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Number of subjects with at least 1 dose-limiting toxicity (DLT) | 28 days post-completion of RT
Number of subjects experiencing treatment-emergent adverse events (TEAE), serious TEAEs, TEAEs leading to discontinuation of RT, and TEAEs leading to death | 28 days post-completion of RT

SECONDARY OUTCOMES:
Identification of dose(s) of XRD-0394 that achieve concentrations within protocol-specified range | Day 2 of RT regimen
Determination of maximum plasma concentration (Cmax) after a single dose of XRD-0394 | Day 2 through Day 5 of RT regimen
Determination of plasma concentrations at 1 to 4 hours post-dose after a single dose of XRD-0394 | Day 2 through Day 5 of RT regimen
Determination of time to maximum plasma concentration (tmax) after a single dose of XRD-0394 | Day 2 through Day 5 of RT regimen
Determination of area under the plasma concentration versus time curve from zero to the last sampling time (AUC0-t) after a single dose of XRD-0394 | Day 2 through Day 5 of RT regimen
Determination of area under the plasma concentration versus time curve from zero to infinity (AUC0-∞) after a single dose of XRD-0394 | Day 2 through Day 5 of RT regimen
Determination of terminal half-life (t1/2) after a single dose of XRD-0394 | Day 2 through Day 5 of RT regimen
Change in radiation-induced phosphorylated Krüppel-associated box domain (KRAB)-associated protein 1 (pKAP1) in tumor biopsy samples | Day 1 through Day 5 of RT regimen

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford Clinical Cancer Center, Stanford, California
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No